CLINICAL TRIAL: NCT06150521
Title: Hysteroscopic Myomectomy for Submucosal Myomas Without Energy Instruments
Status: Active, not recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: K2023084
Record Dates: First submitted 2023-10-12; First posted 2023-11-29 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hysteroscopic Myomectomy
Keywords: Hysteroscopy; Cold knife; Myomectomy; Submucous myoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The hysteroscopic myomectomy group: Patients underwent cold knife hysteroscopic myomectomy

SUMMARY:
Uterine fibroid are the most common benign tumor in the female reproductive system. Although many patients with uterine fibroid do not need to be treated because they are asymptomatic, some patients can experience compression, menorrhagia, pain, irregular bleeding or infertility. The symptoms caused by uterine fibroid are related to its location and size. Submucous fibroids constitute 5-10% of all uterine fibroids.The submucous hysteromyoma is the most likely to cause symptoms, often leads to menorrhagia, irregular bleeding or infertility.

Hysteroscopic myomectomy is a commonly used minimally invasive procedure. The submucous myoma can be resected out by endoscopic resectoscope with electricloop (unipolar and bipolar) . It can preserve the uterus and fertility, also effectively alleviate symptoms.

However, some specific complications have also followed，such as： hemorrhage，uterine perforation， pneumonedema，infections，adhesions，etc. Uterine perforation occurs when the electrode is working, there is a high risk of injury to adjacent anatomical structures. And even without perforation, sometimes thermal injury to adjacent organs may still be discovered in a few days after surgery.In addition，Many scholars have found that hysteroscopic electromyectomy has a higher risk of intrauterine adhesion than other intrauterine operations.

In order to reduce the damage caused by energy source, especially the adverse effects of thermal damage on the endometrium, the new methods of hysteroscopic myomectomy currently include: the hysteroscopic tissue removal (HTR) system, the cold loop myomectomy， the Hysteroscopy Endo Operative system (HEOS)，etc. Existing studies show that，These manipulation techniques did not cause the myometrium damage by radiofrequency energy source, greatly reducing the risk of postoperative intrauterine adhesions. The cold knife hysteroscopic myomectomy in this study is a series of procedures using cold instruments（mechanically, with scissor, grasping or morcellation） to remove uterine submucosal fibroids. The purpose of this surgical technique is to make the operation safe and effective, with greater emphasis on the anatomical and physiological integrity of the myometrial and endometrial layers. This study aims to evaluate the safety and efficacy of cold knife hysteroscopic myomectomy.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria，collecting the data of participants who have undergone cold knife hysteroscopic myomectomy. The investigators will analyze the safety and efficacy of cold knife hysteroscopic myomectomy through the collected data.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent cold knife hysteroscopic myomectomy and excised tissue that showed pathology confirmation of leiomyoma.

Exclusion Criteria:

Patients has gynecologic malignancy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who met the inclusion criteria and underwent cold knife hysteroscopic myomectomy in our hospital being included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Success rate | On the 1 day of surgery
  Total removal of intrauterine pathology with cold knife hysteroscopic myomectomy was defined as a successful operation. During the operation, whether the fibroids were successfully removed by B-ultrasound examination and naked eye
failure rate | On the 1 day of surgery
  Using the cold knife method failed to remove the fibroids. During operative transfer to other surgical methods to remove submucosal fibroids, such as electrical cutting
Incidence of complications | On the 1 day of surgery and on 1 day after surgery
  hemorrhage, pneumonedema, or perforation were registered
surgical bleeding | On the 1 day of surgery and on 1 day after surgery
  Through the intraoperative blood loss assessment and preoperative and postoperative hemoglobin comparison
Checklist of symptom relief | followed-up at 3, 6，12，24 months after surgery
  postoperative menstrual volume, menstrual period, anemia, postoperative fertility, postoperative intrauterine adhesions.

CONTACTS AND LOCATIONS:
Overall Officials: Wanwan Xu, Doctor, Study Chair — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Xu Wanwan, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No